CLINICAL TRIAL: NCT07184489
Title: Validation of the Effectiveness of the CFIR - ERIC Matching Tool in Implementation Research of Pediatric Venous Access Device Selection
Brief Title: Validation of the Effectiveness of the CFIR - ERIC Matching Tool in Implementation Research
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHFudanU0814
Record Dates: First submitted 2025-08-25; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Infusions, Intravenous; Implementation Science
Keywords: implementation strategy; CFIR-ERIC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CFIR-ERIC group (Experimental): Develop implementation strategies for applying evidence to clinical practice using CFIR - ERIC matching tool.
  Interventions: Other: implementation strategies

INTERVENTIONS:
Other: implementation strategies — 1. Analysis of barrier factors: A focus group interview will be conducted. Purposive sampling was used to include senior nurses in the ward, members of the evidence-based group, and doctors for the analysis of barrier factors. Then the CFIR-ERIC matching tool will be used to develop implementation strategies based on the barrier factors.
  2. The best - worst scaling method will be used to generate relatively reliable and valid preference evidence of stakeholders for implementation strategies from CFIR-ERIC matching tool.
  3. The implementation strategies will be developed specifically by an expert group. This group includes nursing managers and experts in evidence-based practice.
  4. Implement the strategies.
  Other Names: pediatric venous access device selection decision tree

SUMMARY:
The goal of this implementation study is to learn if the CFIR-ERIC matching tool is effective indeveloping implementation strategies for pediatric nurse. The evidence practised in this study is the pediatric venous access device selection decision tree from clinical practice guideline on infusion therapy in children. The main questions it aims to answer are:

1. Does the implementation strategies developed by CFIR-ERIC matching tool improve nurses knowledge in venous access devices selection.
2. Does the implementation strategies developed by CFIR-ERIC matching tool lower the error rate of appropriate venous access device selection.

Researchers will compare the CFIR-ERIC group to a blank group to see if CIFR-ERIC matching tool works to improve nurses knowleged and lower the error rate of venous access device selection.

Participants will:

1. Receive the implementation strategies made by CFIR-ERIC matching tool.
2. Using the pediatric venous access device selection decision trees in daily catheterization.
3. Record their venous access device selection informantion, consumables usage and pediatric patients' outcome.

DETAILED DESCRIPTION:
Currently，the evidence-based practice research often isolates barrier assessment from implementation strategy development. At tne same time, many implementation science models being overly complex for clinicians. In Chinese, certain studies still neglect barrier assessment, demonstrate inconsistent conceptualization of implementation strategies, and rarely classify developed strategies.

As a tool for matching and selecting implementation strategies, the CFIR - ERIC matching tool has the characteristics of strong pertinence, repeatability, structuring, systematization, and simple and convenient operation compared with other models. Researchers can identify barrier factors through CFIR and use the CFIR - ERIC matching tool to match strategies to promote the implementation of clinical intervention measures.

This implementation study adopted a pre-post design using the CFIR-ERIC Matching Tool to analyze barriers and develop strategies. Grounded in the "Pediatric Venous Access Device Selection Decision Tree" from the 2021 clinical practice guideline on infusion therapy in children, the intervention was rolled out across 21 wards at the Children's Hospital of Fudan University.

The implementation process of the evidence was evaluated from four aspects using the RE-AIM framework , including the evaluation indicators corresponding to each dimension of patient reach, intervention efficacy, medical adoption, and guideline implementation.

ELIGIBILITY:
Inclusion Criteria:

* Having worked at the research site for ≥ 1 year;
* Being able to independently perform nursing operations (having completed the content related to intravenous infusion in the standardized training of this hospital and passed the assessment).

Exclusion Criteria:

* Not having obtained the nurse practice license;
* Refusing to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
error rate of appropriate venous access device selection | 6 months
  According to the recommendations in the guidelines, selecting the infusion device is considered correct, while failing to select according to the recommendations is considered incorrect. Error rate = Number of incorrect selections / Total number of catheter insertions by nurses

SECONDARY OUTCOMES:
Score of nurses' knowledge questionaire of venous access device selection | The third and sixth months of the research.
  The knowledge questionnaire is divided into three dimensions: device-related knowledge, access-related knowledge, and selection-related knowledge, with a total score of 100. The higher the score, the better the nurses' mastery of knowledge about venous device selection. The online knowledge questionnaire will be distributed to nurses before and after the intervention, and nurses are required to finish it during the morning shift handover. The researchers will conduct statistics on the questionnaire scores.
Nurses' compliance with evidence-based practice behaviors | 6 months
  Develop review indicators based on the evidence from applications, and review whether nurses have achieved the corresponding indicators in clinical practice.
Complication rate | 6 months
  Statistically analyze the incidence of catheter-related complications in children after nurses select intravenous infusion devices.
The cost of venous access device consumables | 6 months
  Including venous access device (including the total number of catheters consumed by successful or failed placement), dressing, central venous maintenance kits, infusion connectors, and flushing or locking solution.
Implementing process evaluated based on "Reach*Efficacy(RE)-Adoption, Implementation, and Maintenance(AIM)" framework | 6 months
  Including Reach, Efficacy, Adoption, Implementation, and Maintenance. Reach refers to the participation rate of training course; Efficacy refers to the change of knowledge level and compliance of evidence-based practice behavior of nurses in the intervention group; Adoption refers to the proportion of evidence actually adopted by nurse in the intervention group and the changes of context; Implementation refers to the completion rate of each training plan in the implementation strategy; Maintenance refers to evaluating the maintenance of the selection scheme.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No